CLINICAL TRIAL: NCT03206125
Title: A Case-Control Study of Esophageal Squamous Cell Carcinoma in Lilongwe, Malawi
Brief Title: NCI UNC Project ESCC
Status: Terminated | Type: Observational
Why Stopped: determined not to be human subjects research
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917120; 17-C-N120
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Case-Control Study; Risk Factors; Epidemiology
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Controls
- ESCC Cases: ESCC Cases

SUMMARY:
Background:

Esophageal cancer is a common cause of cancer deaths. Most cases of this cancer are esophageal squamous cell carcinoma (ESCC). Many of these cases come from two parts of the world with high-risk. One of these is in East Africa and include the country of Malawi. Researchers want to learn what factors explain the high risk there so we can understand better what causes this cancer in people everywhere.

Objective:

To learn more about causes and outcomes of esophageal squamous cell carcinoma using Malawi because of the large number of cases in that country.

Eligibility:

Adults at least 18 years old who have ESCC and live in a certain region of Malawi

Adults in the same age group and location who do not have ESCC

Design:

Participants will be screened at a hospital in Malawi.

Participants will have a 1-hour interview. They will answer questions about:

Demographics (age, ethnicity, education)

Place of residence

Medical history and family medical history

Drug, alcohol, and tobacco use

Hot beverage consumption

Indoor air pollution

Occupation

Food habits

Farming

Gastrointestinal health

Participants will have their teeth and fingernails examined.

Participants will be asked to give samples of blood, urine, saliva, toenails, and for the cancer cases, a small piece of their tumor.

Participants will have 4 phone calls a year for 2 years to ask about their health....

DETAILED DESCRIPTION:
Background: Esophageal cancer causes an estimated 400,000 deaths per year and ranks as the sixth leading cause of cancer death worldwide, just after breast cancer. Esophageal squamous cell carcinoma (ESCC) accounts for 89% of all esophageal cancer cases worldwide and many of the cases originate in two high risk regions, one in Asia and the other in Africa.

Smoking tobacco and heavy alcohol consumption do not explain the incidence rates in the high-risk regions. It is therefore important to consider a wide range of etiologic factors to explain the high rates of cancer in these populations.

Malawi has the highest incidence rates of ESCC in Africa. Our previous studies in Kenya and preliminary studies in Malawi point to a number of potential ESCC risk factors.

Objectives: Our study aims to enhance our understanding of the causes and outcomes for ESCC in Malawi

Eligibility: All suspected ESCC cases will be eligible for enrollment.

Design: We will conduct a case-control study of ESCC jointly at Kamuzu Central Hospital and St. Gabriel s Hospital, recruiting 300 ESCC cases and 300 controls, to (1) evaluate exposures (including consumption of very hot beverages, use of firewood as fuel, tooth loss and animal exposure) which may influence risk of ESCC in Malawi and (2) collect biological samples to quantify exposures of interest (included in the current proposal) and to study the genetics and genomics of ESCC tumors (to be included in a future proposal).

ELIGIBILITY:
* INCLUSION CRITERIA:
* All suspected ESCC cases will be eligible for enrollment.
* All KCH and St Gabriel s patients greater than or eqaul to 18 years of age who are residents of the Central Region of Malawi and are diagnosed with histology-confirmed ESCC will be invited to participate as cases in the study.

EXCLUSION CRITERIA:

* Patients <18 years old
* Those living outside the Central Region, those who are medically unable to complete the study procedures (including questionnaire, biosample collection or endoscopy), and those who are unable to understand the study procedures or give informed consent.

While we do expect to see younger people with ESCC in Malawi (as we have seen in Kenya), cases under the age of 18 are rare: the field team would expect to see one or two a year. This estimate is in line with the cancer registry data from Malawi. Therefore, we will not enroll subjects younger than 18 years old.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 ESCC cases and 300 controls recruited from Kamuzu Central Hospital and St Gabriel s Hospital, Namitete (FWA: 00018517) which is 50 km from Kamuzu Central Hospital located in Lilongwe, Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 648 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Esophageal squamous cell carcinoma | At diagnosis
  Pathology confirmed from endoscopic biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Christian Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- Malawi (2):
  - Kazumu Central Hospital (KCH), Lilongwe
  - St Gabriel's Hospital, Namitete

REFERENCES:
- [Background] White RE, Parker RK, Fitzwater JW, Kasepoi Z, Topazian M. Stents as sole therapy for oesophageal cancer: a prospective analysis of outcomes after placement. Lancet Oncol. 2009 Mar;10(3):240-6. doi: 10.1016/S1470-2045(09)70004-X. Epub 2009 Feb 18. PMID 19230771
- [Background] Liu W, Snell JM, Jeck WR, Hoadley KA, Wilkerson MD, Parker JS, Patel N, Mlombe YB, Mulima G, Liomba NG, Wolf LL, Shores CG, Gopal S, Sharpless NE. Subtyping sub-Saharan esophageal squamous cell carcinoma by comprehensive molecular analysis. JCI Insight. 2016 Oct 6;1(16):e88755. doi: 10.1172/jci.insight.88755. PMID 27734031
- [Background] Mlombe YB, Rosenberg NE, Wolf LL, Dzamalala CP, Chalulu K, Chisi J, Shaheen NJ, Hosseinipour MC, Shores CG. Environmental risk factors for oesophageal cancer in Malawi: A case-control study. Malawi Med J. 2015 Sep;27(3):88-92. doi: 10.4314/mmj.v27i3.3. PMID 26715952